CLINICAL TRIAL: NCT06410300
Title: A Multi-Center Pilot Biomarker Study With Cardiopulmonary Monitoring in Lung Cancer Patients Receiving Combined Thoracic Radiotherapy and Immunotherapy
Brief Title: Cardiopulmonary Monitoring in Lung Cancer Patients Receiving Combined Thoracic Radiotherapy and Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: Bo Lu (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Bo Lu, Chair & Professor, Department of Radiation Oncology, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Other Study IDs: 2093626
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma & PBMC samples will be collected as per protocol required. Samples will be analyzed per protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: Curative Radiotherapy — Radiation dose of 45 Gy or higher
Drug: Immunotherapy — checkpoint inhibitor per PI discretion

SUMMARY:
The overall purpose of this study is to evaluate cardiopulmonary toxicity in patients with lung cancer (NSCLC or SCLC) undergoing combined thoracic radiotherapy ± chemotherapy and immunotherapy through timed monitoring and blood sample collection and to identify correlative biomarkers for predicting cardiopulmonary adverse events.

DETAILED DESCRIPTION:
This aims to collect observational data that describe clinical (primary endpoint) and subclinical (secondary endpoint) cardiopulmonary toxicities from combined thoracic radiotherapy and immunotherapy up to 25 months after thoracic radiotherapy and 12 months after consolidation immunotherapy among patients with locally advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years age
* Diagnosis of locally advanced lung cancer (NSCLC or SCLC) with planned curative radiotherapy (45Gy and above) and planned consolidation immunotherapy.

  * Patients who are not receiving concurrent chemotherapy and radiotherapy are eligible.
  * Patients on a clinical trial that includes thoracic radiotherapy and immunotherapy are eligible and may be co-enrolled to this study.
* ECOG performance status of 0-2
* Life expectancy of 6 months or longer
* Patient able to provide a written informed consent prior to study entry

Exclusion Criteria:

* Prior thoracic radiotherapy to chest.
* Patients are excluded if they are not candidates for curative thoracic radiotherapy or immunotherapy.
* Other severe acute or chronic medical or psychiatric condition that may increase the risk associated with study participation, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 125 patients (MU: 25 patients, UR: 50 patients, Rutgers: 50 patients) who are 18 year of age or older, diagnosed with locally advanced lung cancer (defined as above) will be accrued in the study.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2028-04-19 (Estimated); Study Completion 2030-04-19 (Estimated)

PRIMARY OUTCOMES:
Clinical cardiopulmonary toxicities | 25 months
  To determine clinical cardiopulmonary toxicities from standard RT and immunotherapy per CTCAEv5.0

SECONDARY OUTCOMES:
subclinical/asymptomatic cardiopulmonary events | 25 months
  Asymptomatic cardiopulmonary events determined per abnormal lab values such as troponin and physiological testing

CONTACTS AND LOCATIONS:
Overall Officials: Bo Lu, MD, Principal Investigator — Chair, Department of Radiation Oncology
Locations (3):
- United States (3):
  - University of Missouri - Ellis Fischel Cancer Center, Columbia, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Rochester Medical Center, Rochester, New York